CLINICAL TRIAL: NCT00249223
Title: Risperidone Depot (Microspheres) vs. Risperidone Tablets - a Non-inferiority, Efficacy Trial in Subjects With Schizophrenia
Brief Title: A Comparison of the Effectiveness and Safety of Injectable Risperidone With That of Risperidone Tablets in the Treatment of Patients With Chronic Schizophrenia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Pharmaceutica N.V., Belgium (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR006061
Record Dates: First submitted 2005-11-04; First posted 2005-11-07 (Estimated); Last update posted 2011-01-14 (Estimated); Status verified 2011-01

CONDITIONS: Schizophrenia; Psychotic Disorders
Keywords: chronic schizophrenia, psychotic disorder, risperidone, long-acting injectable, intramuscular injection, antipsychotic agents
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

INTERVENTIONS:
Drug: Risperidone Long acting injectable

SUMMARY:
The primary purpose of the study is to show that treatment with an injectable formulation of risperidone is not less effective than and has a similar safety profile to risperidone tablets in patients with chronic schizophrenia.

DETAILED DESCRIPTION:
Chronic schizophrenia is a longer-term condition that is characterized by a lack of drive, underactivity and slowness, and social withdrawal. As with the acute form of schizophrenia, delusions and hallucinations are common. Based on the severity and long-term nature of this disease, it is important that patients take their antipsychotic medication regularly. Long-acting injectable forms of antipsychotic drugs may eliminate the need for daily oral medication and increase a patient's compliance in taking their medication as prescribed by their physician. This is a randomized, double-blind, parallel-group study comparing the effectiveness and safety of an injectable formulation of risperidone (coated microspheres) to risperidone tablets in patients with chronic, stable schizophrenia. The study is composed of a screening visit, followed by two study phases: an 8-week run-in period and a 12-week double-blind period. In the run-in phase, patients discontinue from other antipsychotic drugs, begin receiving oral risperidone, and stay on the optimal oral risperidone dose that is determined for each patient for 4 weeks before starting the double-blind period. Patients are then randomized to either risperidone tablets or the injectable risperidone formulation at the dose level established during the last 4 weeks of run-in. For the next 12 weeks patients receive an injection of risperidone every 2 weeks plus daily oral doses of placebo or receive a placebo injection every 2 weeks plus daily oral doses of resperidone tablets. The primary measure of effectiveness is the change from baseline in the total score for the Positive and Negative Syndrome Scale for Schizophrenia (PANSS), a rating scale that measures the symptoms of schizophrenia. Additional efficacy testing includes the Clinical Global Impressions (CGI), a rating system used to evaluate the severity of clinical change in a patient with various diseases affecting the brain. Safety evaluations include the incidence of adverse events, results of clinical laboratory tests (hematology, biochemistry, urinalysis), measurements of vital signs and body weight, physical examination and electrocardiogram (ECG) findings, clinical examination of the injection area (buttocks), and the Extrapyramidal Symptoms Rating Scale (ESRS), a scale used to measure effects of antipsychotic medications on motor functions of the patient. The study hypothesis is that the injectable formulation of risperidone will not be less effective than oral risperidone tablets. The injectable formulation of risperidone will be considered less effective than oral risperidone if the improvement in total PANSS with injectable risperidone is more than 6 points worse than the improvement with oral risperidone. Risperidone injections (25, 50 or 75milligrams [mg]) starting Day 1 of the double-blind phase, then every 2 weeks (total of 12 weeks) or 2, 4, or 6mg/day risperidone tablets, starting Day 1 of the run-in period and continuing for the rest of the study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia according to the Diagnostic and Statistical Manual of Mental Diseases, 4th edition (DSM-IV) criteria
* total score on the PANSS at study entry of >=50
* before trial entry, results of clinical hematology, biochemistry, and urinalysis tests performed at screening visit are within normal ranges
* women of child-bearing age must use adequate birth control methods, have a negative pregnancy test before the start of risperidone treatment, and not be breast feeding
* patients' schizophrenia symptoms are stable for the last 4 weeks of the run-in period.

Exclusion Criteria:

* Patients with a DSM-IV Axis I diagnosis other than schizophrenia
* documented disease of the central nervous system that can interfere with the trial assessments, for example stroke, tumor, Parkinson's Disease, Alzheimer's Disease
* moderate or severe symptoms at screening of tardive dyskinesia, a condition of uncontrollable movements of the tongue, lips, face, trunk, hands and feet that is seen in patients receiving long-term medication with certain types of antipsychotic drugs
* history of neuroleptic malignant syndrome, a rare condition in patients receiving antipsychotic medication in which patients may develop fever, sweating, unstable blood pressure, rigid muscles, and other symptoms, including changes in their normal mental state
* acute, unstable or other significant and untreated medical conditions, such as infections, unstable diabetes, or unstable hypertension.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 641 (Actual)
Dates: Start 2000-01; Study Completion 2000-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline to end of double-blind treatment in the total score for PANSS.

SECONDARY OUTCOMES:
CGI Severity Scale; safety evaluations conducted throughout the study.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutica N.V. Clinical Trial, Study Director — Janssen Pharmaceutica N.V.

REFERENCES:
- [Result] Chue P, Eerdekens M, Augustyns I, Lachaux B, Molcan P, Eriksson L, Pretorius H, David AS. Comparative efficacy and safety of long-acting risperidone and risperidone oral tablets. Eur Neuropsychopharmacol. 2005 Jan;15(1):111-7. doi: 10.1016/j.euroneuro.2004.07.003. PMID 15572280